CLINICAL TRIAL: NCT03562312
Title: Clinical, Neuroendocrine and Physiological Effects of Exercise in Patients With Music Performance Anxiety
Brief Title: Performance Anxiety Changes With Exercise
Acronym: PACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Friede Springer Stiftung, Germany (Unknown)
Responsible Party: Principal Investigator, Dr. Jens Plag, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA114217
Record Dates: First submitted 2018-05-03; First posted 2018-06-19 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Performance Anxiety
Keywords: MPA; Music Performance Anxiety; HIIT; Exercise; Cortisol; HRV; Heart Rate
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-intensive aerobe exercise (Experimental): Aerobe bicycle ergometer training within 77-95% of maximum oxygen consumption; duration of each training session: 20 minutes; frequency of training: 6 sessions within 12 days
  Interventions: Other: high-intensive aerobe exercise
- low-intensive aerobe exercise (Placebo Comparator): Aerobe training below 70% of maximum oxygen consumption (including light stretching and simple exercises adapted from yoga figures); duration of training session: 20 minutes; frequency of training: 6 sessions within 12 days
  Interventions: Other: low-intensive aerobe exercise

INTERVENTIONS:
Other: high-intensive aerobe exercise — Aerobe bicycle ergometer training within 77-95% of maximum oxygen consumption; duration of each training session: 20 minutes; frequency of training: 6 sessions within 12 days
  Arms: high-intensive aerobe exercise
Other: low-intensive aerobe exercise — Aerobe training below 70% of maximum oxygen consumption (including light stretching and simple exercises adapted from yoga figures); duration of training session: 20 minutes; frequency of training: 6 sessions within 12 days
  Arms: low-intensive aerobe exercise

SUMMARY:
This study investigates the effect of high-intense aerobe exercise training (HIIT) and aerobe exercise of low intensity on clinical and physiological parameters (anxiety, activity, cortisol, alpha amylase, heart rate, heart rate variability, spiroergometry) in patients with Music Performance Anxiety (MPA). Half of the patients will receive HIIT, while the other half will receive aerobe exercise of low intensity.

DETAILED DESCRIPTION:
In this study, 20 patients with MPA will receive a high-intensive aerobe training (HIIT, 6 HIIT-sessions of 20 minutes within a period of 12 days). Additionally, 20 MPA-patients will undergo a less intense aerobe training matched regarding frequency and duration of sessions. Prior to the first training session, after completing the training (day 12) and 10 days after the Training (day 22), symptoms of anxiety and will be assessed by using questionnaires. Moreover, heart rate and heart rate variability will be obtained and activity level is measured using accelerometers. Before and after the training there will be an assessment of saliva samples for measuring cortisol and alpha amylase.

Furthermore, a standardized performance situation is established before and after the Training. Before, during and after the performance anxiety ratings, cortisol, alpha amylase, heart rate and heart rate variability are assessed.

The investigators hypothesize, that patients with MPA which undergo HIIT, will show a stronger and more sustained improvement of both, clinical symptoms and physiological measures. Specifically, a decreased heart rate, higher heart rate variability and decreased endocrinological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of social anxiety disorder, Performance only subtype due to DSM-5
* Appropriate abilities to communicate and to complete the questionnaires
* Written informed consent
* Possibility of regular attendance at the training sessions
* Participant is a classical instrumentalist

Exclusion Criteria:

* Other severe mental conditions than MPA (e.g. schizophrenia, severe depressive episode, addiction)
* Acute suicidality
* Epilepsy or other disorders of the central nervous system (e.g. tumor, encephalitis)
* Contraindications to aerobe exercise Training
* Start or modification of an anxiolytic pharmacotherapy or other therapy within the last four weeks
* Current psychotherapy
* no sufficient capability to consent to trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-04-14 (Actual)

PRIMARY OUTCOMES:
Bühnenangstfragebogen | Change from Baseline to post therapy (+12 days) and from Baseline to follow-up (+22 days)
  Bühnenangstfragebogen is a questionnaire measuring Music Performance Anxiety. It is the German Version of the PAQ (Performance Anxiety Questionnaire)

SECONDARY OUTCOMES:
Screening für somatoforme Störungen (SOMS-7T) | Change from Baseline to post therapy (+12 days) and from Baseline to follow-up (+22 days)
  SOMS-7T is a questionnaire for detecting the changes in somatisation
Screening für somatoforme Störungen (SOMS-2) | Only one assessment at baseline to assess differences between the two intervention groups
  SOMS-2 is a questionnaire for detecting the severity of somatisation
NEO-FFI personality inventory | Only one assessment at baseline to assess differences between the two intervention groups
  personality inventory measuring neuroticism, extraversion, openness to experience, agreeableness, conscientiousness
Resilienzskala (RS-13) | Change from Baseline to post therapy (+12 days) and from Baseline to follow-up (+22 days)
  A Questionnaire measuring resilience
Trierer Inventar zum chronischen Stress (TICS) | Only one assessment at baseline to assess differences between the two intervention groups
  TICS is an inventory measuring chronic stress
Angstkontrollfragebogen (AKF) | Change from Baseline to post therapy (+12 days) and from Baseline to follow-up (+22 days)
  AKF is the German Version of the Anxiety Control Questionnaire
Anxiety Sensitivity Index (ASI) | Change from Baseline to post therapy (+12 days) and from Baseline to follow-up (+22 days)
  ASI is a Questionnaire measuring anxiety sensitivity
Beck Anxiety Inventory (BAI) | Change from Baseline to post therapy (+12 days) and from Baseline to follow-up (+22 days)
  BAI is a questionnaire measuring anxiety
Beck Depression Inventory (BDI) | Change from Baseline to post therapy (+12 days) and from Baseline to follow-up (+22 days)
  BDI is a questionnaire measuring depression
Liebowitz Social Anxiety Scale (LSAS) | Change from Baseline to post therapy (+12 days) and from Baseline to follow-up (+22 days)
  LSAS is a questionnaire measuring social anxiety
Fragebogen zu sozialphobischen Kognitionen (SPK) | Change from Baseline to post therapy (+12 days) and from Baseline to follow-up (+22 days)
  SPK is the German Version of the social cognitions questionnaire. It measures cognitions in social situations
saliva cortisol hormone | Change from Baseline to post therapy (+12 days) and in performance situations 1 and 2 (+15 days)
  Cortisol is an established marker of the psychophysiological stress response and obtained with help of Salivettes absorbing saliva
saliva alpha Amylase hormone | From Baseline to post therapy (+12 days) and during performance situations 1 (Baseline) and 2 (+15 days)
  Alpha amylase is an established marker of the psychophysiological stress Response and obtained with help of Salivettes absorbing saliva
heart rate | Change from Baseline to post therapy (+12 days), from Baseline to Follow-up and during performance situations 1 (Baseline) and 2 (+15 days)
  Measurement of heart rate
heart rate variability | Change from Baseline to post therapy (+12 days), from Baseline to follow-up (+22 days) and during performance situations 1 (Baseline) and 2 (+15 days)
  heart rate variability is a non-invasive method to measure autonomic nervous System function
visual analogue scale for anxiety (VAS) | Change during performance situations 1 (baseline) and 2 (+15 days)
  VAS is a scale measuring an individual's anxiety in a specific situation
Accelerometer | Change from Baseline to post therapy (+12 days) and from Baseline to follow-up (+22 days)
  With help of an accelerometer the activity level of a person can be measured
International Physical Activity Questionnaire (IPAQ-SF) | Change from Baseline to post therapy (+12 days) and from Baseline to follow-up (+22 days)
  With the IPAQ-SF the physical activity of an individual during the last 7 days can be measured
K-MPAI | Change from Baseline to post therapy (+12 days) and from Baseline to follow-up (+22 days)
  Kenny Music Performance Anxiety Inventory is a questionnaire measuring Music Performance Anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Schmidt, Study Chair — Charite University, Berlin, Germany
Locations (1):
- Department of Psychiatry and Psychotherapy, Charité - Universitätsmedizin Berlin, Campus Mitte, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided